CLINICAL TRIAL: NCT02175238
Title: Relative Bioavailability of BI 691751 Administered With and Without Food to Healthy Male Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1334.28
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BI 691751 after high fat breakfast (Experimental): single dose BI 691751 after a standardised high fat breakfast
  Interventions: Drug: BI 691751 after high fat breakfast
- BI 691751 fasted (Active Comparator): single dose BI 691751 in fasted state
  Interventions: Drug: BI 691751 fasted

INTERVENTIONS:
Drug: BI 691751 fasted — single dose BI 691751 in fasted state
  Arms: BI 691751 fasted
Drug: BI 691751 after high fat breakfast — single dose BI 691751 after a standardised high fat breakfast
  Arms: BI 691751 after high fat breakfast

SUMMARY:
The primary objective of this trial is to investigate the relative bioavailability and pharmacokinetics in plasma and whole blood of BI 691751 administered as a single dose with and without food in healthy male subjects.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the investigator's assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogramm (ECG), and clinical laboratory tests
2. Age 18 to 50 years (incl.)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)

Exclusion criteria:

1. Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and 12-lead Electrocardiogramm (ECG)) deviating from normal and judged clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the study drug
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma and whole blood over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 480 hours
Maximum measured concentration of the analyte in plasma and whole blood (Cmax) | up to 480 hours

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma and whole blood over the time interval from 0 extrapolated to infinity (AUC0-inf) | up to 480 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1334.28.01001 Boehringer Ingelheim Investigational Site, Madison, Wisconsin, United States